CLINICAL TRIAL: NCT06555406
Title: Time-restricted Eating as an Adjunctive Intervention for Bipolar Disorder
Brief Title: Healthy Lifestyles in Bipolar Disorder: Bay Area Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Salk Institute for Biological Studies (Other); University College, London (Other); Swinburne University of Technology (Other); Deakin University (Other); University of British Columbia (Other); Wellcome Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRE_Study2
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Bipolar Disorder; Time Restricted Eating
Keywords: sleep; insomnia; circadian rhythms
MeSH Terms: conditions — Bipolar Disorder; Intermittent Fasting; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: All participants will be assigned to time-restricted eating. Adherence levels are expected to predict change in outcomes and proposed mechanisms. Key hypothesized mechanisms include salivary dim-light melatonin onset and buccal swab assessment of circadian clock genes to assess the amplitude of clock gene expression.
Masking Description: Outcomes will be assessed by interviewers. Where possible, interviewers will be unaware of the treatment condition (interviewers will evaluate symptoms for more than one study, allowing us to keep them unaware of treatment condition).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Time Restricted Eating (TRE) for 8 weeks (Experimental): Participants will receive an intro to TRE and then throughout 8 weeks they will receive brief online psychoeducation several times per week with optional weekly coaching sessions. TRE involves restricting the window of eating to 10 hours/ day, most typically by avoiding eating in the first 1-2 hours after awakening and in the 2-4 before sleep. Those with an eating window > 14 hours will be asked to restrict their eating to 12 hours in the first week, then 10 hours in week 2. To select the period, investigators will ask Ss to review baseline logs to consider sleep, eating, family meals and social commitment schedules, and any special energy demands, such as exercise. During the eating window, no restrictions are placed on the type or quantity of food consumed. The investigators will instruct participants to follow their habitual diet within their 10-hour eating window and to aim to consume the same number of calories per day as they did at baseline.
  Interventions: Behavioral: Time-restricted eating for 8 weeks

INTERVENTIONS:
Behavioral: Time-restricted eating for 8 weeks — limiting food intake to 10 hours per day
  Other Names: intermittent fasting

SUMMARY:
The goal of this clinical trial is to understand how level of adherence with time-restricted eating (TRE) predicts change in diurnal rhythms (as measured using the amplitude of diurnal peripheral clock gene expression), and how those changes predict lower mania and depressive symptoms, and downstream improvements in quality of life. The effects of diurnal amplitude of clock gene expression is expected to remain significant when controlling for change in glucose tolerance and inflammation. Participants will be enrolled who are already receiving medication treatment for bipolar disorder. Participants will complete daily measures of eating, sleep and mood for two weeks, and then will be assigned to follow TRE for eight weeks. Symptoms and Quality of Life will be measured at baseline and during and after the food plan.

DETAILED DESCRIPTION:
This is a single-arm trial to examine the effects of time-restricted eating on change in diurnal rhythms, manic and depressive symptoms, and quality of life. In time-restricted eating (TRE), participants will be asked to limit their food intake to a period of 10 hours per day. TRE will be an addition to standard medication approaches in bipolar disorder. Participants who are receiving medical treatment for bipolar disorder and who report at least some sleep or circadian problems will complete baseline measures and then will be asked to follow TRE for 8 weeks, and then will complete measures of symptoms, Quality of Life, and possible treatment mechanisms at the mid-point of treatment, the end of treatment, and at 3 months after the intervention. If successful, this work will help understand key mechanisms through which TRE provides benefits for those with BD.

ELIGIBILITY:
Inclusion Criteria:

* Meets diagnostic criteria for bipolar I disorder or bipolar II disorder (but not cyclothymia, bipolar disorder Not otherwise specified or bipolar disorder due to another medical condition) assessed by the Diagnostic Interview for Anxiety, Mood, and Obsessive-compulsive and Related Neuropsychiatric Disorders [DIAMOND])
* current sleep (insomnia, hypersomnolence) or circadian sleep-wake (delayed phase, advanced phase, irregular sleep-wake, non-24-hour sleep-wake-type) concerns indicated by endorsement of at least some sleep or circadian-related impairment across the screening self-reports or interview
* Living in an English-speaking country (and one that the researchers have expertise in research procedures and diet)
* Has been speaking English for at least 10 years, speaks English in the home, or certifies that they are able to understand English well for the study and demonstrates this during the screening interview.
* Receiving medical care for bipolar disorder (referrals will be provided for those who would like to begin care)
* Mood-stabilizing medication regimens stable for at least one month
* < 5 kg weight change in the past 3 months
* Currently eating ≥ 12 hours per day at least twice per week
* Able to operate the camera function and respond to web-based surveys by phone (loaner phones will be provided as needed)
* Not engaged in current shift work or have other responsibilities such as providing care that would chronically disrupt their sleep (i.e., > 3 h between 22:00 and 05:00 h for at least 1 day/week)
* Able to complete 7 days of dietary logs adequately (e.g., at least 2 entries per day, covering at least a 5-hour eating window) during the baseline period
* Able to complete screening and baseline questionnaires adequately (e.g., not failing more than 1 attention check item with instructed responding; responding to standard multiple-choice items in a mean of < 2 seconds per item). Where individuals respond to more than 14 items in a row with the same response, their answers will be manually reviewed for possible invalidity.

Exclusion criteria include the following:

* Current episode of depression, hypomania or mania, or psychosis (assessed by the DIAMOND), Participants with acute mood disorder episodes will be encouraged to seek treatment and to consider the study when symptoms have remitted.
* Eating disorder diagnosis (by self-report of treatment or diagnosis at any point during their life, Short Eating Disorder Examination Questionnaire (EDE-QS) scores above clinical concern thresholds for eating disorders, or DIAMOND interview of symptoms during adulthood)
* Past 3-month alcohol use disorder or substance use disorder (assessed by DIAMOND)
* Active suicidal ideation coupled with plan, intent or attempt history as assessed by Columbia Suicide Severity Rating Scale
* Conditions that would interfere with ability to take part in the intervention, including pregnancy, breastfeeding, uncorrected hypo or hyperthyroidism, gastrointestinal conditions impairing nutrient absorption
* Conditions that would confound immune or other study measures, such as HIV, AIDS, lupus, or multiple sclerosis
* Medications contraindicated for fasting: clozapine, glucose-lowering medications, diabetes-related injections, medications requiring food early morning or late evening, corticosteroids; Glucagon-like peptide-1 (GLP-1) agonists will not be an exclusion criteria if weight stabilized
* Cognitive deficits as noted during the initial interview or as indicated by low performance on the Orientation Memory Concentration Test- Short Version (weighted score < 20)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Mania | Lower YMRS at the end of intervention (10 weeks) as compared to baseline
  Young Mania Rating Scale (YMRS) total scores (minimum: 0, maximum: 60, high scores reflect higher manic symptom severity)
Depression | Lower MADRS at the end of intervention (10 weeks) as compared to baseline
  Montgomery Asberg Depression Scale (MADRS) total scores (minimum: 0, maximum: 60, higher scores reflect higher depressive symptom severity)
Self-rated Quality of Life (QOL) | Scores at 1.5-months post-intervention (16 weeks) as compared to baseline
  self-rated Brief Quality of Life in Bipolar Disorder (QoL.BD) (minimum: 12, maximum: 60, higher scores reflect better QOL)

SECONDARY OUTCOMES:
Mania at follow-up | YMRS and LIFE scores will be lower at 3 months post-intervention as compared to baseline
  YMRS (described above) and Longitudinal Interval Follow-up Evaluation (LIFE; minimum 0, maximum 6) scores across follow-up (higher scores reflect more severe symptoms)
Depression at follow-up | MADRS scores will be lower at 3 months post-intervention as compared to baseline
  MADRS scores (described above) across follow-up
Self-rated mania | Lower PMQ scores at post-intervention (10 weeks) and at 1.5 and 3 months follow-ups post-intervention, as compared to baseline
  Patient Health Questionnaire (PMQ) Mania scores (minimum: 0, maximum: 27, higher scores reflect more severe mania)
Self-rated depression | post-intervention (10 weeks) and at 1.5 and 3 months follow-ups post-intervention, as compared to baseline
  Patient Health Questionnaire (PHQ) Depression scores (minimum: 0, maximum: 27, higher scores reflect more severe depression)
Acceptability | immediately post-treatment (10 weeks after enrollment)
  Participant self-ratings of the acceptability of the intervention: The primary index of acceptability will be the percentage of individuals who endorse that they agree or strongly agree that they would recommend the food plan to a friend. This single item has been used in previous trials of bipolar disorder. Higher agreement will be considered a positive outcome.
Weekly change in mania severity | Weekly scores from the end of the intervention through 3 months post-intervention
  Longitudinal Interval Follow-up Evaluation (LIFE) weekly mania scores post-treatment as compared to those at baseline. The investigators will administer the LIFE interview at 6 months after study entry, and interviewers will record a mania severity rating for each week, to cover the time from the end of intervention until 6-month follow-up. Better outcomes would be reflected in lower LIFE scores post-treatment.
Daily emotional lability as assessed using ecological momentary assessment | 7 weeks post-study entry as compared to baseline
  Mean square of successive difference of negative affect scores within derived from the ecological momentary assessments at 7 weeks post-baseline as compared to baseline. Participants will be asked to complete negative affect ratings 5 times per day for 7 days, at the baseline and mid-point of treatment. The investigators will calculate scores to examine the degree of negative affect variability for each day, and then take the average across 7 days at baseline and at treatment mid-point. Better outcomes would be indicated by lower scores.

CONTACTS AND LOCATIONS:
Overall Officials: Sheri L Johnson, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Measures, data, and analysis scripts will be shared through Open Science Foundation.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: De-identified data will be shared within one year after data collection ends.
Access Criteria: Data will be available publically through Open Science Foundation upon request. Wellcome Trust guidance for data sharing will be followed.

REFERENCES:
- [Derived] Johnson SL, Murray G, Manoogian ENC, Mason L, Allen JD, Berk M, Panda S, Rajgopal NA, Gibson JC, Bower CD, Berle EF, Joyner K, Villanueva R, Michalak EE, Kriegsfeld LJ. A pre-post trial to examine biological mechanisms of the effects of time-restricted eating on symptoms and quality of life in bipolar disorder. BMC Psychiatry. 2024 Oct 21;24(1):711. doi: 10.1186/s12888-024-06157-5. PMID 39434066